CLINICAL TRIAL: NCT00107471
Title: A Phase I/II Study of Topotecan With G-CSF and Radiation Therapy in Children With Malignant Intrinsic Pontine Brainstem Gliomas of Childhood
Brief Title: Topotecan, G-CSF, and Radiation Therapy in Treating Young Patients With Newly Diagnosed Brain Stem Glioma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The unpromising experience of the French group with topotecan given at a dosage of 0.4 mg/m2/day over 30 mins w/in 1 hr of radiation (Cancer 2005; 104: 2792).
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACNS0224; CDR0000417842 (Other: Clinical Trials.gov); COG-ACNS0224 (Other: Children's Oncology Group)
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Brain Tumors; Central Nervous System Tumors
Keywords: untreated childhood brain stem glioma
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Topotecan; Radiotherapy; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose Level I (0.5 mg/m^2) (Experimental): Radiation Therapy + Topotecan hydrochloride daily before each dose of irradiation (radiation therapy) + filgrastim (G-CSF) (p.r.n)
  Interventions: Biological: filgrastim; Drug: topotecan hydrochloride; Radiation: radiation therapy
- Dose Level 2 (0.6 mg/m^2) (Experimental): Radiation Therapy + Topotecan hydrochloride daily before each dose of irradiation (radiation therapy) + filgrastim (G-CSF) (p.r.n.)
  Interventions: Biological: filgrastim; Drug: topotecan hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim — Given PO
  Other Names: Granulocyte Colony-Stimulating Factor; r-metHuG-CSF; G-CSF; Neupogen; NSC #614629
Drug: topotecan hydrochloride — Given IV
  Other Names: SKF-104864; Hycamtin; NSC #609699
Radiation: radiation therapy
  Other Names: Conformal therapy or Intensity modulated radiation therapy (IMRT) may be; used.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Colony-stimulating factors, such as G-CSF, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Radiation therapy uses high-energy x-rays to kill tumor cells. Topotecan may make tumor cells more sensitive to radiation therapy . Giving topotecan and G-CSF together with radiation therapy may be an effective treatment for brain stem glioma.

PURPOSE: This phase I/II trial is studying the side effects and best dose of topotecan when given together with G-CSF and radiation therapy and to see how well they work in treating young patients with newly diagnosed brain stem glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of escalating the dose of topotecan when administered with filgrastim (G-CSF) and radiotherapy, in terms of increasing the topotecan dose 25-50% above the maximum tolerated dose (MTD) determined in a prior phase I study, in young patients with newly diagnosed malignant intrinsic pontine brain stem glioma. (Phase I)
* Determine the dose-limiting toxic effects of topotecan in these patients. (Phase I)
* Determine the 1-year event-free survival and overall survival of patients treated with this regimen (at the MTD of topotecan determined in phase I). (Phase II)
* Determine the toxicity of this regimen in these patients. (Phase II)

Secondary

* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a multicenter, phase I, dose-escalation study of topotecan followed by a phase II study.

* Phase I: Patients receive topotecan IV over 30 minutes followed by radiotherapy once daily, 5 days a week for 6-7 weeks. During chemoradiotherapy, patients also receive filgrastim (G-CSF) IV or subcutaneously daily, if needed, until blood counts recover. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 out of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive topotecan (at the MTD determined in phase I ), G-CSF, and radiotherapy as in phase I.

After completion of study treatment, patients are followed within 2 weeks, every 3 months for 1.5 years, every 6 months for 1.5 years, and then annually until disease relapse.

PROJECTED ACCRUAL: A total of 3-72 patients (3-12 for phase I and 60 for phase II) will be accrued for this study within approximately 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of intrinsic pontine brain stem glioma within the past 30 days

  * Histologic confirmation not required provided the tumor has a pontine epicenter AND exhibits diffuse (rather than focal) involvement of ≥ 2/3 of the pons with or without extension to the adjacent medulla or midbrain* NOTE: *Brain stem tumors that do not meet these criteria must be histologically confirmed as grade III or IV malignant glioma
* Measurable disease by radiographic imaging

  * Post-operative MRI required within the past 30 days if patient had a biopsy or surgical resection
* No disseminated disease
* No neurofibromatosis type 1

PATIENT CHARACTERISTICS:

Age

* 3 to 21 at diagnosis

Performance status

* Lansky 50-100% OR
* Karnofsky 50-100%

Life expectancy

* At least 8 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3 (transfusion independent)
* Hemoglobin ≥ 10.0 g/dL (transfusion allowed)

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT < 2.5 times ULN

Renal

* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR
* Creatinine based on age as follows:

  * No greater than 0.8 mg/dL (for patients ≤ 5 years of age)
  * No greater than 1.0 mg/dL (for patients 6 to 10 years of age)
  * No greater than 1.2 mg/dL (for patients 11 to 15 years of age)
  * No greater than 1.5 mg/dL (for patients over 15 years of age)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Not severely somnolent or comatose

  * Central cortical neurotoxicity scale < grade 3

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunomodulating agents

Chemotherapy

* No other concurrent anticancer chemotherapy

Endocrine therapy

* Concurrent corticosteroids allowed for neurological deficits related to the tumor

Radiotherapy

* No prior radiotherapy

Surgery

* See Disease Characteristics
* Prior biopsy or surgical resection for malignant brain stem glioma allowed

Other

* No other prior therapy for malignant brain stem glioma

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2005-10; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure (e.g., tumor progression, tumor recurrence, or death from any cause) | From date of enrollment until the first occurrence of relapse, progressive disease, secondary malignancy, or death or until last contact if none of these events occur, assessed up to 3 years

SECONDARY OUTCOMES:
Time to death | From the time of study entry to the first occurrence of death by any cause

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L. Robertson, MD, Study Chair — University of Michigan Rogel Cancer Center; Richard A. Axtell, MD, Study Chair — Helen DeVos Children's Hospital at Spectrum Health
Locations (80):
- United States (72):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama-Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Cancer Center, Sacramento, California
  - Stanford Comprehensive Cancer Center - Stanford, Stanford, California
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - University of Illinois Cancer Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Kosair Children's Hospital, Louisville, Kentucky
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center & Children's Hospital - Fairview, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth - Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (3):
  - Royal Children's Hospital, Herston, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (4):
  - Children's Hospital of Western Ontario, London, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
- Swiss Pediatric Oncology Group Bern, Bern, Switzerland